CLINICAL TRIAL: NCT05685420
Title: Extension Study of Herombopag in Children and Adolescents With Chronic Primary Immune Thrombocytopenia
Brief Title: Extension Study of Herombopag for Pediatric Patients With Chronic Immune Thrombocytopenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-TPO-ITP-III-PED-EXT
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: open-label Herombopag plus standard of care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open-label (Experimental): Herombopag plus standard of care
  Interventions: Drug: Herombopag

INTERVENTIONS:
Drug: Herombopag — Thrombopoietin receptor agonist

SUMMARY:
The main purpose of this extended study is to enable subjects who are currently receiving the PartB experimental drug in the HR-TPO-ITP-III-PED clinical trial .To continue receiving the experimental drug after the completion of the clinical trial if they benefit from the treatment at the end of the clinical trial.Until the study physician determines that the subject has failed treatment or that the subject can no longer benefit from treatment or extends the study treatment for 6 months.In addition, the secondary purpose of this extended study was to observe the long-term efficacy and safety of tripodal in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed PartB of HR-TPO-ITP-III-PED clinical trial and have achieved platelet response.
2. Subjects who have signed the informed consent for the extended study.
3. Subjects with potential fertility（e.g. women who have menarche or men who have sperm loss) should agree to use effective contraception during their participation in the extended study and within 28 days after their last dose.
4. Subjects who have completed end-of-treatment visits in the original study.

Exclusion Criteria:

1. Any unstable condition or condition that may compromise the safety of the subject.
2. Patients with new myelofibrosis were examined in the original clinical trial exit group.
3. The original clinical trial cohort examined evidence of new cataract or existing cataract progression, and the study considered it unsuitable to enroll in this extension.
4. Patients with uncontrolled bleeding after standard treatment.
5. Any previous occurrence of arterial or venous thrombosis (transient ischemic attack,myocardial infarction ,deep venous thrombus, or pulmonary embolism ),or clinical symptoms and history suggest thrombus susceptibility.
6. Any other circumstances that the investigator considers likely to cause the subject to be unable to complete the study or to present a significant risk to the subject.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Estimated)
Dates: Start 2023-01-23 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with new myelofibrosis，new cataract, or existing cataract progression during the extended study. | from baseline to 28 days after the last dose
All AESIs，whether or not associated with study drugs. | from baseline to 28 days after the last dose
All SAEs，whether or not associated with study drugs. | from baseline to 28 days after the last dose
All AEs that result in discontinuation of medication. | from baseline to 28 days after the last dose
All AEs that lead to permanent withdrawal. | from baseline to 28 days after the last dose
Blood Biochemistry-ALT. | 6 months
Blood Biochemistry-AST. | 6 months
Blood Biochemistry-GGT. | 6 months
Blood Biochemistry-ALP. | 6 months
Blood Biochemistry-TBIL. | 6 months
Blood Biochemistry-DBIL. | 6 months
Blood Biochemistry-creatinine. | 6 months

SECONDARY OUTCOMES:
Platelet count at each visiting point. | 6 months
The incidence and severity of bleeding symptoms. | 6 months
  According to the 2021 version go pediatric ITP bleeding Score Scale.
Percentage of subjects receiving emergency treatment for aggravated ITP. | 6 months
Percentage of subjects with recurrent ITP. | 6 months

IPD SHARING:
Plan to Share IPD: Undecided